CLINICAL TRIAL: NCT02939170
Title: Initial Performance of a Daily Disposable Contact Lens Featuring Molded Marks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLO870-C001
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-12

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DT1 MF MM (Experimental): Delefilcon A multifocal contact lenses with molded marks on back surface worn bilaterally (in both eyes) for 9 hours
  Interventions: Device: Delefilcon A Multifocal Contact Lenses with Molded Mark
- DT1 MF (Active Comparator): Delefilcon A multifocal contact lenses worn bilaterally for 9 hours
  Interventions: Device: Delefilcon A Multifocal Contact Lenses

INTERVENTIONS:
Device: Delefilcon A Multifocal Contact Lenses with Molded Mark
  Arms: DT1 MF MM
Device: Delefilcon A Multifocal Contact Lenses
  Other Names: DAILIES TOTAL1® Multifocal (DT1 MF)
  Arms: DT1 MF

SUMMARY:
The purpose of this study is to evaluate the impact of back surface molded marks (MM) applied to delefilcon A contact lenses as measured by the incidence of ocular discomfort device-related adverse events with DAILIES TOTAL1® Multifocal contact lenses with molded marks (DT1 MF MM) and current DAILIES TOTAL1® Multifocal contact lenses (DT1 MF).

ELIGIBILITY:
Inclusion Criteria:

* Must sign an Informed Consent document;
* Current wearer of commercial DAILIES TOTAL1® contact lenses;
* Have spectacles in current prescription available to be worn in conjunction with the investigational product;
* Manifest astigmatism less than or equal to 0.75 diopter (D) (at screening)
* Best corrected distance visual acuity (BCVA) greater than or equal to 20/25 in each eye;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Eye injury in either eye within 12 weeks prior to study enrollment;
* Any anterior segment infection, inflammation, disease, or abnormality that contraindicates contact lens wear;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated;
* History of herpetic keratitis, refractive surgery or irregular cornea;
* A pathologically dry eye that precludes contact lens wear;
* Concurrent participation in a contact lens or contact lens care product clinical trial within the previous 30 days;
* Monocular (only 1 eye with functional vision);
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2016-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, CTM, Study Director — Alcon, A Novartis Division
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 study centers located in the United States.
Pre-assignment Details: Of the 87 enrolled, 7 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (80).
Period: Overall Study
Arm/Group | DT1 MF MM | DT1 MF
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any study lenses (Safety Analysis Set).
Groups:
- DT1 MF MM: Delefilcon A multifocal contact lenses with molded marks on back surface worn bilaterally for 9 hours
- Total: Total of all reporting groups
Arm/Group | DT1 MF MM | DT1 MF | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.47) | 36.1 (10.07) | 36.2 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Ocular Discomfort Device-related Adverse Events (AE)
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device (test article). Ocular discomfort device-related AE was defined as an ocular AE classified as "Related" to study device and deemed to be related to ocular discomfort.
Time Frame: Day 1 at Hour 9
Population: Safety Analysis Set
Measure: Number; unit: Events
Units Other Than Participants: Eyes
Arm/Group | DT1 MF MM | DT1 MF
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 80 | 80
Events | 0 | 1

2. Secondary Outcome: Ocular Staining
Description: Assessed by the Investigator through slit-lamp examination and graded on a 5-point scale, where 0=none and 4=severe. Ocular staining was categorized by corneal staining, conjunctival staining, and limbal staining. Both eyes contributed to the analysis.
Time Frame: Day 1 at Hour 9
Population: Safety Analysis Set
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | DT1 MF MM | DT1 MF
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 80 | 80
Eyes
  Corneal Staining, Grade 0 | 62 | 63
  Corneal Staining, Grade 1 | 14 | 17
  Corneal Staining, Grade 2 | 4 | 0
  Corneal Staining, Grade 3 | 0 | 0
  Corneal Staining, Grade 4 | 0 | 0
  Conjunctival Staining, Grade 0 | 60 | 61
  Conjunctival Staining, Grade 1 | 15 | 15
  Conjunctival Staining, Grade 2 | 5 | 4
  Conjunctival Staining, Grade 3 | 0 | 0
  Conjunctival Staining, Grade 4 | 0 | 0
  Limbal Staining, Grade 0 | 72 | 67
  Limbal Staining, Grade 1 | 7 | 13
  Limbal Staining, Grade 2 | 1 | 0
  Limbal Staining, Grade 3 | 0 | 0
  Limbal Staining, Grade 4 | 0 | 0

3. Secondary Outcome: Limbal Hyperemia
Description: Hyperemia (excess of blood) was assessed by the Investigator through slit-lamp examination and graded on a 5-point scale, where 0=none and 4=severe. Both eyes contributed to the analysis.
Time Frame: Day 1 at Hour 9
Population: Safety Analysis Set
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | DT1 MF MM | DT1 MF
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 80 | 80
Eyes
  Grade 0 | 60 | 52
  Grade 1 | 20 | 27
  Grade 2 | 0 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (1 day). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device (test article). AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to initiation of study treatment
- DT1 MF MM: All subjects exposed to delefilcon A multifocal contact lenses with molded marks
- DT1 MF: All subjects exposed to delefilcon A multifocal contact lenses
Arm/Group | Pre-treatment | DT1 MF MM | DT1 MF
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/87 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.